CLINICAL TRIAL: NCT05116397
Title: Influence of Graded Hypercapnia on Endurance Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: USARIEM
Record Dates: First submitted 2021-10-13; First posted 2021-11-11 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hypercapnia
MeSH Terms: conditions — Hypercapnia

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded crossover design
Who Masked: Participant
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4% CO2 (Experimental): Inspired gas containing 4% CO2, 21% O2, balance N2
  Interventions: Other: Inspired gas
- 2% CO2 (Experimental): Inspired gas containing 2% CO2, 21% O2, balance N2
  Interventions: Other: Inspired gas
- 0% CO2 (Sham Comparator): Inspired gas containing 0% CO2, 21% O2, balance N2
  Interventions: Other: Inspired gas

INTERVENTIONS:
Other: Inspired gas — Inspired gas content

SUMMARY:
The aim of this randomized, single-blind, placebo-controlled crossover trial is to determine the effects of graded hypercapnia (0, 2, and 4% inspired CO2) on endurance performance. Twelve healthy and fit young adults (men and women) will complete this study. Participants will perform experimental trials on 3 separate days (one each breathing 0%, 2%, and 4% inspired CO2-all with normal 21% oxygen). During each trial, they will perform 10 minutes of submaximal treadmill walking exercise and then complete a self-paced 2-mile treadmill run time-trial.

DETAILED DESCRIPTION:
Participants will undergo baseline measurements of pulmonary function and maximal oxygen uptake (VO2max). They will then complete two familiarization trials, with 10 minutes of submaximal exercise (~40%VO2max) followed by a self-paced 2-mile treadmill time trial. Lastly, they will complete three experimental trials, repeating the same submaximal and time-trial exercise procedures while breathing the test gas (0%, 2%, or 4% CO2-all with normal 21% oxygen). During the experimental trials, arterialized capillary blood samples will be collected at rest breathing room air, at rest breathing the test gas, and during submaximal exercise at 40% VO2max breathing the test gas. The primary outcome is 2-mile treadmill time-trial performance. Secondary outcomes include ventilation, metabolic rate, heart rate, arterialized capillary pH/PCO2/HCO3, perceived exertion, dyspnea, leg discomfort, breathing descriptors, and headache ratings.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-45
* In good health as determined by medical screening
* Passed his/her most recent Army Combat Fitness Test (ACFT) (Military Volunteers Only) or performs aerobic exercise at least 2 times per week and able to complete two mile run in ≤ 21 minutes (Civilian Volunteers)
* Willing to not participate in any exercise or drink alcoholic beverages for 24 hours before each study visit.
* Willing to not take part in any strenuous exercise in the 36 hours before each visit.
* Willing not to drink caffeine or eat food until after testing on familiarization and performance testing visits (visits 2-6).
* Willing to maintain a similar dietary pattern in the 2 days before each familiarization and performance visits.
* Have supervisor approval if permanent party military or a federal employee at U.S. Army Natick Soldier System Center
* Able to speak and read English fluently

Exclusion Criteria:

* Females who are pregnant or planning to become pregnant during the study
* Taking dietary supplements, prescriptions, or over the counter medication, other than a contraceptive (unless approved by medical staff & PI)
* Musculoskeletal injuries that compromise ability to run on a treadmill
* Abnormal blood count, presence of abnormal blood chemicals (hemoglobin S or sickle cell traits)
* Smokers or tobacco/nicotine users (unless have quit > 1 month prior)
* Any history of asthma
* Current or recent respiratory tract or sinus infections (< 1 month prior)
* Allergy to skin adhesive
* Any history of migraine or recurrent headaches
* Any history of panic disorder
* Blood donation in the previous 8 weeks
* Positive Covid-19 test within the last month

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
2 mile self-paced treadmill time trial performance | 30 minutes
  Time to complete self-paced 2 mile treadmill time trial (min:sec)

SECONDARY OUTCOMES:
Ventilation rate | 30 minutes
  Ventilation rate will be assessed using a pneumotachometer [L/min]
Oxygen consumption | 30 minutes
  Oxygen consumption will be assessed using computerized indirect calorimetry [ml/kg/min]
Heart rate | 30 minutes
  Heart rate will be assessed using telemetry [beats per min]
Arterialized capillary pH | 30 minutes
  Arterialized capillary pH will be assessed using a blood gas analyzer [Unitless]
Arterialized capillary pCO2 | 30 minutes
  Arterialized capillary pCO2 will be assessed using a blood gas analyzer [mmHg]
Arterialized capillary HCO3 | 30 minutes
  Arterialized capillary HCO3 will be assessed using a blood gas analyzer [mEq/L]
Rating of perceived exertion | 30 minutes
  Rating of perceived exertion will be assessed using Borg's 6-20 scale [AU]
Dyspnea | 30 minutes
  Rating of perceived dyspnea will be assessed using Borg's 0-10 scale [AU]
Leg discomfort | 30 minutes
  Rating of perceived leg discomfort will be assessed using Borg's 0-10 scale [AU]
Headache | 30 minutes
  Headache will be assessed using a visual analog scale [AU]
Breathing descriptors | 30 minutes
  Breathing descriptors will be assessed by having participants check statements that apply to their breathing (e.g., breathing out requires more effort) [unitless]

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Ryan, Ph.D., Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT05116397/ICF_000.pdf